CLINICAL TRIAL: NCT02912104
Title: A Therapeutic Trial of Human Amniotic Epithelial Cells Transplantation for Primary Ovarian Failure
Acronym: POF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Principal Investigator, Dongmei Lai, Principal Investigator, International Peace Maternity and Child Health Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20152236
Record Dates: First submitted 2016-09-06; First posted 2016-09-23 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Primary Ovarian Insufficiency; Premature Ovarian Failure; Infertility
Keywords: primary ovarian insufficiency; premature ovarian failure; Infertility; human amniotic epithelial cells transplantation
MeSH Terms: conditions — Primary Ovarian Insufficiency; Infertility | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hAECs transplantation (Experimental): To clarify the safety and effectiveness of human amniotic epithelial cells transplantation for the treatment of POF patients
  Interventions: Biological: human amniotic epithelial cells (hAECs) transplantation

INTERVENTIONS:
Biological: human amniotic epithelial cells (hAECs) transplantation — hAECs are prepared and cultured using GMP(Good Manufacturing Practice, GMP) rules, 3×10^7 hAECs in 4.5ml is separately injected into ovarian tissue by bilateral ovarian artery infusion.
  Other Names: hAECs transplantation

SUMMARY:
This project will clarify the safety and effectiveness of human amniotic epithelial cells transplantation for the treatment of primary ovarian failure (POF) patients and provide a new therapeutic method for patients with infertility.

DETAILED DESCRIPTION:
POF is a defect characterized by the premature depletion of ovarian follicles. Patients with POF suffer from amenorrhea, infertility, low levels of estrogen, and high gonadotropin concentration before the age of 40. The early failure of ovarian function leads to lost fertility and increases risk of osteoporosis and cardiovascular disease, which has serious impact on the patient's physical, mental health and family stability. The etiology of POF is complex, and so far there has not been any effective treatment. Recent study showed that human amniotic epithelial cells (hAECs), also known as the birth waste, are newly discovered adult stem cells. The hAECs have the ability to repair nerve damage, myocardial injury, as well as liver damage. hAECs have low immunogenicity and no ethical restrictions. Therefore, hAECs are expected to become the new seed cells for regenerative medicine. Our previous study was the first to show that human amniotic epithelial cells have the ability to restore folliculogenesis in a mouse model with chemotherapy-induced premature ovarian failure. Our further studies demonstrated that hAECs either directly transdifferentiated into granulosa cells, or inhibited tumor necrosis factor-alpha-mediated granulosa cell apoptosis and reduced the inflammatory reaction in ovaries induced by chemotherapeutics, regulating VEGFA and its receptors to induce follicular growth related to paracrine activity. Therefore, it is necessary to start the clinical study of human amniotic epithelial cells transplantation in the POF disease which may offer a novel therapeutic strategy for improving the quality of life of POF patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and<45 years old.
2. Female patients with documented diagnosis of POF: <40 years old, at least 4 months of amenorrhea not due to pregnancy, two FSH levels above 40 IU/L, at least one month apart.
3. Not in other trial within 3 months prior to the start of this trial.
4. Willing to participate in this trial and to give informed consent/assent before any procedures are performed in this trial.

Exclusion Criteria:

1. History of, or evidence of current malignancy within the past 5 years.
2. Severe functional impairment of vital organs.
3. Abnormal karyotype.
4. Coagulation disorders.
5. Severe pelvic adhesions.
6. Uncontrolled acute or chronic gynecologic inflammation.
7. Congenital adrenal cortical hyperplasia.
8. Cushing's syndrome.
9. Thyroid dysfunction.
10. Pituitary adenoma.
11. Pituitary amenorrhea or Hypothalamic amenorrhea.
12. Thrombophlebitis, venous thrombosis or artery thrombosis.
13. History of Oophorocystectomy.
14. Currently pregnant or breast-feeding.
15. Currently receiving other treatment that might affect the efficacy and safety of stem cells.
16. History of severe drug allergy.
17. Active infection detected by chest X-ray/CT.
18. HIV, TPAb positive.
19. Mental illness.
20. Currently participating in any other clinical trial that uses interventional drugs or examinations.
21. Patients that are deemed, by the investigator, inappropriate to participate in this trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability assessed by Adverse Events | 150 days
  Proportion of patients with adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESI，such as acute allergic reaction, ectopic mass formation related to treatment)

SECONDARY OUTCOMES:
Change from baseline in bilateral ovarian volume | 150 days
  The ovarian volume will be assessed by pelvic ultrasound on 30th, 90th, 150th days after transplantation.
Change from baseline in number of antral follicles (AFC) | 150 days
  The number of antral follicles developing will be assessed by pelvic ultrasound on 30th, 90th, 150th days after transplantation.
Change from baseline in Follicle-stimulating hormone (FSH) serum level | 150 days
  Serum FSH level will be tested on 30th and 150th days after transplantation.
Change from baseline in Luteinizing hormone (LH), Estradiol (E2), Testosterone (T), Prolactin (PRL) , Anti-müllerian hormone (AMH) serum level | 150 days
  Serum LH, E2, T, PRL, AMH level will be tested on 30th and 150th days after transplantation.
Menstruation resumption | 150 days
  Patients will monitor for resumption of menses within 150 days after transplantation. If the menstruation resumption rate is over 30%, the treatment will be considered effective.
Endometrial thickness | 150 days
  The endometrial thickness will be assessed by pelvic ultrasound on 30th, 90th, 150th days after transplantation.
Bone mineral density (BMD) measurements | 150 days
  The BMD will be tested on 150th day after transplantation.
Achievement of pregnancy | 12 Months
  Achievement of pregnancy by natural or assisted conception methods, such as in vitro fertilization (IVF). The outcomes of pregnancy include conception, miscarriage and delivery.
  If the pregnancy rate is over 30%, the treatment will be considered effective.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Lai, M.D., Principal Investigator — The center of Laboratory, The international peace Maternity and child health Hospital,School of Medicine, Shanghai Jiaotong University, Shanghai,China,200030
Locations (1):
- The International Peace Maternity and Child Health Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The public can require the data and protocol from clinicaltrials.gov posted by investigator
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: public
URL: https://clinicaltrials.gov

REFERENCES:
- [Result] Wang F, Wang L, Yao X, Lai D, Guo L. Human amniotic epithelial cells can differentiate into granulosa cells and restore folliculogenesis in a mouse model of chemotherapy-induced premature ovarian failure. Stem Cell Res Ther. 2013 Oct 14;4(5):124. doi: 10.1186/scrt335. PMID 24406076
- [Result] Zhang Q, Xu M, Yao X, Li T, Wang Q, Lai D. Human amniotic epithelial cells inhibit granulosa cell apoptosis induced by chemotherapy and restore the fertility. Stem Cell Res Ther. 2015 Aug 25;6(1):152. doi: 10.1186/s13287-015-0148-4. PMID 26303743
- [Result] Yao X, Guo Y, Wang Q, Xu M, Zhang Q, Li T, Lai D. The Paracrine Effect of Transplanted Human Amniotic Epithelial Cells on Ovarian Function Improvement in a Mouse Model of Chemotherapy-Induced Primary Ovarian Insufficiency. Stem Cells Int. 2016;2016:4148923. doi: 10.1155/2016/4148923. Epub 2015 Nov 9. PMID 26664408
- [Derived] Weng L, Wei L, Zhang Q, Sun T, Kuang X, Huang Q, Cao Y, Liu X, Wang Q, Guo Y, Sun J, Wang L, Tang H, Yang H, Chen Q, Zhang J, Wang B, Qian Z, Lai D. Safety and efficacy of allogenic human amniotic epithelial cells transplantation via ovarian artery in patients with premature ovarian failure: a single-arm, phase 1 clinical trial. EClinicalMedicine. 2024 Jul 30;74:102744. doi: 10.1016/j.eclinm.2024.102744. eCollection 2024 Aug. PMID 39165278